CLINICAL TRIAL: NCT05628727
Title: Comparison of Intermittent Fasting Interventions on Brain Health in Women: A Randomized Controlled Trial
Brief Title: Intermittent Fasting Interventions on Brain Health in Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting
Sponsor: McMaster University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14969
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5:2 Fasting Group (Experimental): This group will use the 5:2 method and fast for two non-consecutive days of the week.
  Interventions: Other: 5:2 Fasting
- Time-Restricted Feeding Group (Experimental): This group will use the 16:8 method every day, eating only during an 8-hour period that will commence at wake-up time.
  Interventions: Other: Time Restricted Feeding
- Control Group (No Intervention): This group will not fast.

INTERVENTIONS:
Other: Time Restricted Feeding — This group will use the 16:8 method every day, eating only during an 8-hour period that will commence at wake-up time.
  Other Names: TRF
  Arms: Time-Restricted Feeding Group
Other: 5:2 Fasting — This group will use the 5:2 method and fast for two non-consecutive days of the week.
  Other Names: 5:2 Method
  Arms: 5:2 Fasting Group

SUMMARY:
Adults experience high psychological stress due to many factors such as school, workplace, or personal life. Adult women are known to experience higher stress levels than men. Current evidence shows that fasting improves mental health outcomes in men. The research is unclear on fasting interventions and their potential impact on stress levels in women. In this study, investigators will compare two fasting diets over 8 weeks. There will be a control group, one group that fasts for two days per week, and a final group that only eats for 8 hours in the morning. Mental health surveys, brain tests and a blood draw will be done during the study to see any mental or physical changes from the diets. Investigators will study the motivation of women to continue the diet during and beyond the study through online surveys.

ELIGIBILITY:
Inclusion Criteria:

* English speaker
* Assignment of female sex at birth
* BMI between 18.5-24.9 kg/m^2
* Current engagement in less than 150 minutes of physical activity per week
* Normal menstrual cycle length (21-40 days) for at least 3 months
* Non-smoker
* Consumption of no more than one alcoholic beverage per day
* Mild to higher levels of stress as indicated by a score of 15 or higher on the stress sub-set of the DASS-21 questionnaire

Exclusion criteria:

* Pregnant or breastfeeding
* Diagnosed chronic disease (cardiovascular, metabolic, respiratory, reproductive, renal, neuromuscular, or any other disease or condition as assessed by the Canadian Society for Exercise Physiology Get Active Questionnaire)
* Diagnosed eating disorder
* Participation in a weight-loss program in the last 3 months
* Loss of 5% of body weight or more in the last 3 months

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-09-06 (Actual); Study Completion 2025-09-06 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21) Questionnaire - Stress Sub-Scale | 8 weeks
  Investigators will administer the standardized DASS-21 Questionnaire at Week 0 and Week 8. The stress sub-scale will be used to measure any potential effects of fasting interventions on psychological stress over time.
  The scoring of answers is based on a 0 to 3 scale. 3 reflects the negative extreme on the Likert Scale. Scores range from 0-42, higher scores are indicative of higher psychological stress levels.

SECONDARY OUTCOMES:
Colour and Word Stroop Test (SCWT) | 8 weeks
  Investigators will administer the standardized SCWT at Week 0 and Week 8 to assess the potential effects of fasting interventions on selective attention and response inhibition in participants over time.
  This task requires participants to name the displayed colour of the presented words while they disregard the meaning of the words.
  Several outcome measures will be produced:
  1. Reaction time (RT) in milliseconds (ms)
  2. The Stroop Effect - the difference in RT between incongruent and congruent trials, which can be broken down into 2 components:
     1. Stroop interference effect - the RT difference between incongruent and neutral trials
     2. Stroop facilitation effect - the RT difference between the neutral and congruent trials
Mnemonic Similarity Task (MST) | 8 weeks
  Investigators will administer the standardized MST to assess the potential effects of fasting interventions on high interference memory over time.
  Several outcome measures will be produced:
  1. Reaction time
  2. High-interference memory (assessed as the ability to correctly identify lure items as ''Similar'')
  3. General recognition memory performance (assessed as the ability to correctly identify repetitions items as ''Old'')
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  Investigators will administer the standardized PSQI at Week 0 and Week 8 to measure the self-reported quality and patterns of sleep in adults.
  Several outcomes will be measured:
  1. Subjective sleep quality
  2. Sleep latency
  3. Sleep duration
  4. Habitual sleep efficiency
  5. Sleep disturbances
  6. Use of sleeping medication
  7. Daytime dysfunction over the last month
  The scoring of answers is based on a 0 to 3 scale. 3 reflects the negative extreme on the Likert Scale. Scores range from 0-21, where higher scores are indicative of poorer sleep quality and a global score of >5 is indicative of poor sleep quality.
Eating Disorder Examination Questionnaire (EDE-Q 6.0) | 8 weeks
  Investigators will administer the standardized EDEQ-6.0 during screening and Week 8 to measure self-reported disordered eating patterns in adults and the potential effects of fasting interventions on this outcome measure over time.
  2 main outcomes will be measured:
  1. Frequency data on key behavioural features of eating disorders in terms of the number of episodes of the behaviour.
  2. Sub-scale scores reflect the severity of characteristics of eating disorders. The sub-scales are Restraint, Eating Concern, Shape Concern and Weight Concern.
  Generally, sub scales are measures on a 7-point Likert scale. Higher scores on the global scale and sub-scales denote more problematic eating behaviours and attitudes.
Profile of Mood States (POMS) | 8 weeks
  Investigators will administer the standardized POMS at Week 0 and Week 8 to measure the potential effects of fasting interventions on self-reported quality and patterns of sleep in adults over time.
  Several outcomes will be measured:
  1. Total Mood Disturbance [TMD] (-32 to 200)
     Subscales:
  2. Anger (0-48)
  3. Confusion (0-28)
  4. Depression (0-60)
  5. Fatigue (0-28)
  6. Tension (0-36)
  7. Vigour (0-32)
  The scoring of answers is based on a 5-point Likert scale (not at all - extremely). Higher TMD scores are indicative of a poorer mood state.
State Anxiety Inventory (STAI) Short Form | 8 weeks
  Investigators will administer the standardized STAI at Week 0 and Week 8 to measure the potential effects of fasting interventions on self-reported state and trait anxiety levels over time.
  All items are rated on a 4-point Likert scale (e.g., from "Almost Never" to "Almost Always"), with higher scores indicating greater anxiety levels.
Five Facet Mindfulness Questionnaire (FFMQ) | 8 weeks
  Investigators will administer the standardized FFMQ at Week 0 and Week 8 to measure the potential effects of fasting interventions on the self-reported trait-like tendency to be mindful in daily life. It is comprised of the following five related facets: observing, describing, acting with awareness, non-judging, and non-reactivity.
  The 39 items of the FFMQ are rated on a 5-point Likert scale: ranging from 1 (never or very rarely true) to 5 (very often or always true). Facet scores can also be combined to produce an overall mindfulness score.
  A higher score indicates a greater trait-like tendency to be mindful in daily life.
Blood Pressure | 8 weeks
  Investigators will use an automated sphygmomanometer to measure blood pressure during each of the 2 in-lab sessions.
  Several measures will be collected:
  1. MAP (mmHg)
  2. Systolic pressure (mmHg)
  3. Diastolic pressure (mmHg)
Height (cm) | 8 weeks
  Investigators will use a vertical scale via measuring tape to measure height (cm) during each of the 2 in-lab sessions.
Weight (kg) | 8 weeks
  Investigators will use an automated scale to measure weight (kg) during each of the 2 in-lab sessions.
Waist Circumference (cm) | 8 weeks
  Investigators will use a flexible measuring tape to measure waist circumference (cm) during each of the 2 in-lab sessions.
Inflammatory Biomarker Interleukin-6 [IL6] (pg/mL) | 8 weeks
  A trained researcher who has completed phlebotomy course will take ~8 ml of blood will be drawn from an antecubital (forearm) vein at rest. The blood will be used to measure biomarkers of inflammation (e.g., proinflammatory cytokines IL6, TNF-a, CRP) during 2 in-lab sessions at week 0 and week 8.
  Measures will be recorded in pg/mL. A higher value will indicate higher levels of inflammation.
Inflammatory Biomarker Tumour Necrosis Factor Alpha [TNF-a] (pg/mL) | 8 weeks
  A trained researcher who has completed a phlebotomy course will take ~8 ml of blood will be drawn from an antecubital (forearm) vein at rest. The blood will be used to measure biomarkers of inflammation (e.g., proinflammatory cytokines IL6, TNF-a, CRP) during 2 in-lab sessions at week 0 and week 8.
  Measures will be recorded in pg/mL. A higher value will indicate higher levels of inflammation.
Inflammatory Biomarker C-Reactive Protein [CRP] (mg/L) | 8 weeks
  A trained researcher who has completed a phlebotomy course will take ~8 ml of blood will be drawn from an antecubital (forearm) vein at rest. The blood will be used to measure biomarkers of inflammation (e.g., proinflammatory cytokines IL6, TNF-a, CRP) during 2 in-lab sessions at week 0 and week 8.
  Measures will be recorded in mg/L. A higher value will indicate higher levels of inflammation.
Blood Ketone Levels (mmol/L) | 8 weeks
  Participants will perform finger pricks using a lancing device and measure blood ketone levels using a ketometer. Values will be recorded in mmol/L, with higher values indicating higher levels of circulating blood ketones.
Blood Glucose Levels (mmol/L) | 8 weeks
  Participants will perform finger pricks using a lancing device and measure blood ketone levels using a glucometer. Values will be recorded in mmol/L, with higher values indicating higher levels of circulating blood glucose.
Body Composition (% Body Fat) | 8 weeks
  Body composition (% body fat and lean body mass) will be measured in participants by investigators using a DEXA (DXA) scanner during the 2 in-lab sessions at Week 0 and Week 8. Higher percentages indicate a higher percent body fat and lower relative lean body mass.
Body Composition (Lean Body Mass - kg) | 8 weeks
  Body composition (% body fat and lean body mass) will be measured in participants by investigators using a DEXA (DXA) scanner during the 2 in-lab sessions at Week 0 and Week 8. Measures will be recorded in kg. A higher lean body mass indicates a lower relative body fat percentage.
Body Mass Index (BMI) | 8 weeks
  Body Mass Index will use participant height and weight as input values to produce a measure in kg/m^2 at Week 0 and Week 8. A higher BMI score indicates a relatively higher body fat percentage.
Diet Satisfaction & Adherence Questionnaire | 8 weeks
  Investigators will administer standardized questions taken from the Diet Satisfaction Questionnaire in addition to adherence questions to measure weekly dietary satisfaction and adherence to the fasting interventions during the intervention.
  Scoring is qualitative.
Pregnancy Status | One time measure at Week 0
  Investigators will collect a urine sample and test it to determine the pregnancy status of the participant as per the exclusion criteria.
  A test strip will be placed in the urine. A positive pregnancy status will be indicated by the appearance of 2 lines in their respective locations on the strip. A negative pregnancy status will be indicated by the presence of only one line in its respective location on the strip.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Heisz, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada